CLINICAL TRIAL: NCT02002637
Title: Evaluation of the Latella Implant System for Lateralization of the Iliotibial Band to Offload the Medial Condyle for Pain Relief in Patients With Medial Osteoarthritis - A Safety Study
Brief Title: Feasibility of the Latella Implant System for Medial Osteoarthritis (OA)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor election
Sponsor: Cotera, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: COT1-13-01; COTERA-1
Record Dates: First submitted 2013-12-02; First posted 2013-12-06 (Estimated); Last update posted 2017-04-28 (Actual); Status verified 2017-04

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

ARMS (1):
- Latella Knee Implant System (Experimental)
  Interventions: Device: Latella Knee Implant System

INTERVENTIONS:
Device: Latella Knee Implant System

SUMMARY:
The objective of this study is to evaluate the safety and technical feasibility of implanting the Latella Implant System in the treatment of patients with medial osteoarthritis of the knee.

ELIGIBILITY:
Inclusion Criteria:

* History of pain as due to medial osteoarthritis

Exclusion Criteria:

* Rheumatoid arthritis
* Joint or ligament instability
* Metal ion allergy

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2013-11; Primary Completion 2015-09 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Freedom from unanticipated serious adverse device effects | 12 Months

CONTACTS AND LOCATIONS:
Overall Officials: Manoj Ramachandran, MD, Principal Investigator — Barts & The London NHS Trust
Locations (2):
- Slotervaart Hospital, Amsterdam, Netherlands
- Barts Health NHS Trust, London, United Kingdom